CLINICAL TRIAL: NCT03736057
Title: Pharmacogenic Guidance to Optimize Safety and Efficacy of Psychotropic Drug Use in Treatment of Behavioral and Psychiatric Symptoms in Dementia
Brief Title: Genetic Evaluation for Medication Selection (GEMS) Study
Acronym: GEMS
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Geldmacher, Professor of Neurology, University of Alabama at Birmingham
Other Study IDs: IRB-150902001
Record Dates: First submitted 2018-10-09; First posted 2018-11-08 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Dementia; Psychiatric Disorders Mood; Behavior Disorders
MeSH Terms: conditions — Dementia; Mood Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva by cheek swab and/spit cup
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Delayed results of pharmacogenomic results — 1:1 randomization schedule for delayed knowledge of pharmacogenomic results to clinician and patient. Results are released to prescriber at <1 week (unblinded) or 12 weeks (blinded). When genomic results are available upon receipt, unblinded clinicians select an FDA-approved drug from the "recommended" drugs when possible. Blinded prescribers provide the intended prescription when notified of blinded status. At 4 weeks, 1° outcome measures, NPI-Q and side effects ratings are collected. Clinicians make a GO/NO-GO decision for continuation based on those measures. A NO-GO decision is unblinding and an alternative drug may be prescribed. At 12 weeks, 1° outcomes are collected again. Previously blinded clinicians will be unblinded and may decide to continue or revise the treatment plan based on the clinical outcomes and the genetic results. After the 12 week visit, results of the genetic tests will be entered in the EHR. Further clinical follow-up is based on need.

SUMMARY:
Investigators propose to determine whether knowing details about how a person's genes affect the way medicines work in the brain and body will help doctors pick more effective or safer medicine for that person. Target symptoms are restlessness, agitation, depression and related problems common in people with memory loss and dementia.

DETAILED DESCRIPTION:
This project offers an innovative approach to improving treatment outcomes for people with Behavioral and psychiatric symptoms of dementia (BPSD), as well as a novel electronic health record (EHR) -compatible means of assessing treatment response. To date, there has been limited investigation of pharmacogenomic testing among people with dementia. Testing has mostly been focused on testing a single Cytochrome P450 (CYP)polymorphism to guide treatment decisions for cognitive enhancing cholinesterase inhibitor medications in patients with Alzheimer disease. Pharmacogenomic guidance of prescribing decisions for psychotropic medications has not been studied for BPSD but there is growing evidence that such analyses can assist in effective prescription decisions for treatment of depression. Since affective symptoms are among the most prominent drivers of BPSD and associated distress, and the highest level evidence for successful treatment of BPSD is with the antidepressant drug citalopram, investigators believe that pharmacogenomic guidance for selection of drugs to treat BPSD is truly innovative, and will provide new insights on implementing safer and more effective treatment for BPSD.

Additionally, investigators will explore the use of the NIH-sponsored Patient Reported Outcomes measurement Information System (PROMIS) as an outcome measure for BPSD. PROMIS is a system of highly reliable, valid, flexible, precise, and responsive assessment tools that measure patient-reported health status. PROMIS measures are available for typical BPSD like anger, anxiety, and depression, but their utility has not been studied in a sample of dementia patients. They offer the potential, through patient-portal EHR interfaces, for clinicians to track treatment responses in a more timely and efficient manner than traditional clinic-based instruments, placing less burden on patients and families to present for in-clinic assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Score <26 on the Alabama Brief Cognitive screen or <24 on the Montreal Cognitive Assessment.
2. Have a caregiver/informant/family member who spends at least 10 hours per week with the affected person and who is willing to participate
3. Be rated by a caregiver/informant as scoring ≥9 on the Functional Activities Questionnaire, including at least one domain score of 3 (dependent).
4. Have BPSD sufficient for the treating clinician to begin or change psychotropic drugs, and of sufficiently mild severity that a delay of 5 days before changing the prescription would not be harmful to the patient.

Exclusion Criteria:

1. BPSD of sufficient severity or intensity that (in clinician's opinion) require immediate medication change or referral for emergency services
2. Lack of reliable informant with adequate exposure to patient and ability to communicate with study staff in English

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As director of the Division of Memory Disorders, PI Dr. Geldmacher leads the effort of the four neurologists and two nurse practitioners who provide clinical services at the UAB Memory Disorders Clinic (MDC). During 2013, there were 1595 total outpatient MDC visits for patients with dementia-related diagnoses. A sample of 100 consecutive MDC patients from April 2015 demonstrated that 69 were treated with psychotropic agents, including antidepressants (n=67), antipsychotics (n=6), or both.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Psychiatric Symptoms of Dementia | 12 weeks
  Comparison from baseline Neuropsychiatric Inventory-Questionnaire (NPI-Q) and the 12-week follow-up.
  Neuropsychiatric Inventory-Questionnaire is a questionnaire completed by caregivers about patients designed to measure both neuropsychiatric symptoms (e.g., agitation/aggression, anxiety, hallucinations). There are 12 symptoms included in NPI-Q. Each domain includes an initial response of "yes" or "no". If "yes", then the caregiver rates the severity of the symptom on a 3-point scale (1= mild, 2=moderate and 3=severe). The NPI-Q provides a total severity score ranged 0-36 with higher scores indicating more severe symptoms.
Behavioral Symptoms of Dementia | 12 weeks
  Comparison from baseline Patient Reported Outcomes Measurement Information System (PROMIS) and the 12-week follow-up.
  This assessment is a self- or informant-rated measure that ascertains mental health domains that are important across psychiatric diagnoses. The scale is used as screener for symptoms severity of the following domains: Anger, anxiety, depression and sleep disturbance. Each item on the measure is rated on a 5-point scale with higher scores reflect greater symptom severity. A rating of mild (i.e., 2) or greater on any item within a domain may serve as a guide for additional inquiry and follow up to determine if a more detailed assessment for that domain is necessary. On the subscales noted above, The raw scores should be summed to obtain a total raw score and identify the associated T-score
  The T-scores are interpreted as follows:
  Less than 55 = None to slight 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe

CONTACTS AND LOCATIONS:
Overall Officials: David Geldmacher, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided